CLINICAL TRIAL: NCT03532932
Title: International, Multicentre, Non-Interventional Study To Evaluate Disease Control And Treatment Pattern In Patients With Moderate To Severe Inflammatory Bowel Disease In Real Life Practice
Brief Title: A Study to Evaluate Disease Control and Treatment Pattern in Participants With Moderate to Severe Inflammatory Bowel Disease (IBD) in Real Life Practice
Acronym: INTENT
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5005; U1111-1207-6263 (Other: WHO)
Record Dates: First submitted 2018-05-01; First posted 2018-05-22 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-09

CONDITIONS: Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UC Participants: Participants diagnosed with moderate to severe UC from approximately 35 investigational sites will be observed retrospectively for previous 2 years before enrollment until Visit 1 and will be observed prospectively for 1 year after participant's enrollment into the study to assess treatment patterns and treatment outcomes in UC participants particularly on the use of available biological therapies.
- CD Participants: Participants diagnosed with moderate to severe CD from approximately 35 investigational sites will be observed retrospectively for previous 2 years before enrollment until Visit 1 and will be observed prospectively for 1 year after participant's enrollment into the study to assess treatment patterns and treatment outcomes in CD participants particularly on the use of available biological therapies.

SUMMARY:
The purpose of this study is to characterize the treatment patterns associated with biologics agents use or non-biological therapy in participants with moderate to severe Ulcerative Colitis (UC) and Crohn's Disease (CD).

DETAILED DESCRIPTION:
This is a non-interventional, retrospective and prospective study of participants with IBD. This study will collect data to provide accurate and comprehensive information related to treatment patterns associated with biologics use or non-biological therapy in participants with moderate to severe UC and CD in routine clinical practice.

The study will have retrospective data collection from past records of participants within the last 2 years before participant's enrollment. The prospective part of the study will include one year of observation and data collection after the participant's enrollment in the study.

The study will enroll approximately 2000 participants. Participants will be enrolled in one of the two groups:

* UC Participants
* CD Participants

This multi-center trial will be conducted in Russia, Belarus and Kazakhstan. The overall period of observation in this study will be approximately 12 months. Participants will make 2 visits within their routine practice to the clinic after the enrollment into the study including a final visit at Month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Has confirmed diagnosis of CD or UC for at least 2 years prior to enrollment in the study.
2. Has a moderate to severe IBD flare at the time of enrollment or in participant anamnesis within 2 years before enrollment treated with steroids or/ and immunosuppressive agents or/ and biologic therapy. IBD flare(s) must be confirmed in the source documentation.
3. Current treatment with steroids or/ and immunosuppressive agents or/ and 5-aminosalicylate (ASA) or/ and biologic therapy.

Exclusion Criteria:

1. Current or previous (within the last two years) indeterminate or not classified colitis.
2. Changing of IBD type in anamnesis (that is, from UC to CD, etc) within the last two years.
3. Current, previous (within the last two years) or planned (for the next one year) participation in interventional clinical trial.
4. Presenting of mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
5. Has received previous treatment with biologic therapy/immunosuppressive agents for conditions other than IBD ever in their lifetime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with moderate to severe UC or CD will be observed both retrospectively and prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 1990 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (36):
- Belarus (2):
  - Republican Gastroenterology Center, City Clinical Hospital # 10, Minsk, Minsk Oblast
  - Vitebsk regional clinical specialized center, Vitebsk, Vitebsk Oblast
- Kazakhstan (3):
  - Scientific-Research Institute of Cardiology and Internal Diseases, Gastroentorology department, Almaty, Almaty Region
  - The Centre of Coloproctology based at City Hospital 1, Astana, Astana
  - Regional clinical hospital, Shymkent, Shymkent
- Russia (31):
  - Regional Clinical Hospital, Barnaul, Altai Territory
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Health of the Russian Federation, Ufa, Bashkortostan Republic
  - State Budgetary Healthcare Institution "Chelyabinsk Regional Clinical hospital", Chelyabinsk, Chelyabinsk Oblast
  - State Budgetary Healthcare Institution Irkutsk Order of the Badge of Honor Regional Clinical Hospital, Irkutsk, Irkutsk Oblast
  - State Autonomous Healthcare Institution of Kemerovo region "Kemerovo regional clinical hospital n. a. S.V. Belyaev", Kemerovo, Kemerovo Oblast
  - Regional State Budgetary Healthcare Institution "Regional Clinical Hospital # 1 n. a. S.I. Sergeev", Khabarovsk, Khabarovsk Territory
  - Budgetary Institution "Surgut District Clinical Hospital", Surgut, Khanty-Mansi Autonomous Okrug-Yugra
  - State Budgetary Institution "Regional Clinical Hospital No. 1 named after Professor S.V. Ochapovsky"., Krasnodar, Krasnodarskiy Kray
  - Krasnoyarsk Interdistrict Clinical Hospital No. 20 named after IS Berzon, Krasnoyarsk, Krasnoyarsk Region
  - Federal State Budget Military Educational Institution of Higher Education "Military Medical Academy named after S.Kirov" of the Ministry of Defense of the Russian Federation, Saint-Petersburg, Leningradskaya Oblast'
  - Scientific and Research Center "Eco-safety", LLC, Saint-Petersburg, Leningradskaya Oblast'
  - St. Petersburg State Budgetary Healthcare Institution "City Clinical Hospital No. 31", Saint-Petersburg, Leningradskaya Oblast'
  - MEDSI Clinical Hospital, Krasnogorsk, Moscow Oblast
  - Moscow Clinical Scientific Center, Moscow, Moscow Oblast
  - State Scientific Center of Coloproctology, Moscow, Moscow Oblast
  - State Budgetary Healthcare Institution Moscow Regional Research and Clinical Institute (MONIKI) n. a. M. F. Vladimirskiy, Moscow, Moscow Oblast
  - Regional Clinical Hospital, Omsk, Omsk Oblast
  - Perm regional clinical hospital, Perm, Perm Krai
  - Medical Academy n. a. S. I. Georgievksiy Federal State Autonomous Educational Institution of Higher Education "Crimean State University n. a. V.I. Vernadskiy, Simferopol, Republic Crimea
  - State Budgetary Healthcare Institution Republic of Crimea "Republican clinical hospital n.a. N.A.Semashko", Simferopol, Republic Crimea
  - Federal State Budget Educational Institution of Higher Education "Petrozavodsk State University", Petrozavodsk, Republic of Karelia
  - Health Care Unit # 1 of Yoshkar-Ola city, Yoshkar-Ola, Republic of Maruy El
  - State Budgetary Institution of Ryazan Region "City Clinical Hospital #4", Ryazan, Ryazan Oblast
  - Society with limited liability "Medical Association" New Hospital ", Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Hospital Ministry of health Republic of Tatarstan, Kazan', Tatarstan Republic
  - Budgetary Institution of Health in the Republic of Udmurtia First Republican Clinical Hospital under the Ministry of Health, the Republic of Udmurtia, Izhevsk, Udmurtiya Republic
  - State Budgetary Healthcare Institution RB Regional Clinical Hospital G.G Kuvatov, Ufa, Ufa Region
  - State Budgetary Healthcare Institution City Clinical Hospital 21, Ufa, Ufa Region
  - State Healthcare Institution Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast
  - Regional Clinical Hospital, Vladimir, Vladimirskaya Oblast’
  - Federal State Budgetary Educational Institution of Higher Education "Chita state medical academy" of the Ministry of Health of the Russian Federation, Chita, Zabaykalskiy (Transbaikal) Kray

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the 36 investigative sites in Russia, Belarus and Kazakhstan from 20 July 2018 to 08 November 2021.
Pre-assignment Details: Participants diagnosed with moderate to severe Ulcerative Colitis (UC) or Crohn's Disease (CD) were observed retrospectively within 2 years before enrollment and prospectively one year after enrollment. A total of 1990 participants were enrolled (signed informed consent) into the study, of which 89 were screen failures. 1901 participants started the study and were analyzed in the study.
Groups:
- UC Participants: Participants diagnosed with moderate to severe UC were observed retrospectively for previous 2 years before enrollment until Baseline Visit 1 (Day 1) and further observed prospectively for 1 year after participants were enrolled into the study during Observational Visit 2 at 6 months and Final Visit 3 at 12 months to assess treatment patterns and treatment outcomes.
- CD Participants: Participants diagnosed with moderate to severe CD were observed retrospectively for previous 2 years before enrollment until Baseline Visit 1 (Day 1) and further observed prospectively for 1 year after participants were enrolled into the study during Observational Visit 2 at 6 months and Final Visit 3 at 12 months to assess treatment patterns and treatment outcomes.
Period: Overall Study
Arm/Group | UC Participants | CD Participants
Started | 1214 | 687
Completed | 1140 | 615
Not Completed | 74 | 72
Not completed — Protocol Deviation | 33 | 31
Not completed — Appearance of Exclusion Criteria | 9 | 11
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 15 | 9
Not completed — Adverse Event | 4 | 3
Not completed — Death | 0 | 2
Not completed — Other | 11 | 16

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included those participants who signed the informed consent form and were analyzed in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | UC Participants | CD Participants | Total
Number analyzed (Participants) | 1214 | 687 | 1901
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.44 (13.63) | 36.44 (13.90) | 39.63 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 582 | 341 | 923
  Male | 632 | 346 | 978
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Russian | 858 | 574 | 1432
  Tartarian | 133 | 38 | 171
  Ukrainian | 4 | 3 | 7
  Baskirian | 24 | 1 | 25
  Chuvash | 2 | 0 | 2
  Belarusian | 24 | 14 | 38
  Kazakh | 88 | 21 | 109
  Other | 81 | 36 | 117
Region of Enrollment [Count of Participants; unit: Participants]
  Belarus | 30 | 14 | 44
  Kazakhstan | 121 | 30 | 151
  Russia | 1063 | 643 | 1706
Employment Status [Count of Participants; unit: Participants]
  Employed | 702 | 343 | 1045
  Unemployed | 287 | 189 | 476
  Pensioner | 133 | 54 | 187
  Student | 53 | 79 | 132
  Other | 39 | 22 | 61
Disability [Count of Participants; unit: Participants] — Disability was determined based on participant's healthcare resources utilization.
  Participants
    Had Disability | 392 | 341 | 733
    Had no Disability | 822 | 346 | 1168
Smoking Status [Count of Participants; unit: Participants]
  Non-smoker and Never Smoked Before | 937 | 519 | 1456
  Ex-smoker | 211 | 93 | 304
  Current Smoker | 66 | 75 | 141
Age at Disease Onset [Mean (Standard Deviation); unit: years] | 34.46 (13.17) | 30.79 (13.57) | 33.14 (13.43)
Family History of Inflammatory Bowel Disease (IBD) [Count of Participants; unit: Participants] — Participants were stratified by the following categories: with IBD history and without IBD history.
  Participants
    With IBD History | 34 | 21 | 55
    Without IBD History | 1180 | 666 | 1846
Clinical Course of IBD [Count of Participants; unit: Participants]
  Acute Form (Less than 6 months Since the Onset of the Illness) | 13 | 9 | 22
  Chronic Continuous Form (Absence of Remission Longer Than 6 months Despite Adequate Treatment) | 362 | 293 | 655
  Chronic Relapsing Course (With Remission Periods Longer Than 6 months) | 839 | 385 | 1224
Complications of IBD [Count of Participants; unit: Participants]
  Had Complications of IBD | 111 | 317 | 428
  Had no Complications of IBD | 1103 | 370 | 1473
Extraintestinal Manifestation (EIM) [Count of Participants; unit: Participants] — Extraintestinal manifestation means when disease impacts other part of body. Between 25-40 percent (%) of IBD participants experience EIMs, commonly in the joints, skin, bones, eyes, kidneys, and liver.
  Participants | 295 | 229 | 524
Had Medical History [Count of Participants; unit: Participants] | 274 | 178 | 452

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Stratified by Treatment Patterns Associated With Biologics Agents Use or Non-biological Therapy in Participants With Moderate to Severe UC and CD
Description: Treatment pattern with biologics agents or non-biological therapy included unique treatments combinations, Like>5-ASA1(Start with 5-ASA:5-ASA→Systemic biologics [SB] +/- STER+/-standard therapy[ST]),>5ASA2(without [w/o] STER),>5ASA3(5-ASA→STER+/-ST),>5ASA4(5-ASA→IS),>5ASA 5(5-ASA→5-ASA+/-IS),>5ASA6(5-ASA→ NOTR),>5ASA7(5-ASA),>NOTR1(NOTR→Biologics [BIO]+/-ST+/-STER),>NOTR 2(TR→ST+/-STER),>NOTR 3(NOTR),>IS1(IS→SB+STER+/-ST),>IS2(IS→SB+ST w/o STER),>IS 3(IS→STER+/-ST),>IS4(IS→5-ASA),>IS5(IS→NOTR),>IS6(IS→5-ASA+IS),>IS7(IS mono),>IS+5ASA1(IS+5-ASA→SB +/-ST),>IS+5ASA2(IS+5-ASA→SB ±ST w/o STER),>IS+5ASA3(IS+5-ASA→STER+/-ST),>IS+5ASA4(IS+5-ASA→NOTR),>IS+5ASA5(IS+5-ASA→IS),>IS+5ASA6(IS+5-ASA→5-ASA),>IS+5ASA7(IS+5-ASA),>BIO1(SB+/-STER+/-ST→withdrawal [w/d] of SB+ST+/-STER),>BIO2(SB+/-STER+/-ST),>BIO3(SB+/-STER+/-ST→NOTR),>BIO4(SB+/-STER+/-ST→SB mono),>STER1(STER+/-ST→w/d of STER+SB+/-ST),>STER2(STER+/-ST→w/d of STER+ST),>STER3(STER+/-ST→SB+STER+/-ST),>STER4(STER+/-ST→NOTR),>STER5(STER+/-ST).
Time Frame: From 2 years before enrollment up to Month 12 after enrollment (up to 3 years)
Population: FAS included those participants who signed the informed consent form and were analyzed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1214 | 687
Participants
  Greater than (>) 5-aminosalicylic acid (5ASA) 1 | 33 | 16
  >5ASA 2 | 38 | 14
  > 5ASA 3 | 192 | 30
  >5ASA 4 | 9 | 5
  >5ASA 5 | 46 | 7
  >5ASA 6 | 22 | 8
  >5ASA 7 | 73 | 5
  >BIO 1 | 28 | 20
  >BIO 2 | 71 | 96
  >BIO 3 | 7 | 22
  >BIO 4 | 9 | 19
  >Immunosuppressive (IS) 1 | 2 | 13
  >IS 2 | 6 | 20
  >IS 3 | 3 | 6
  >IS 4 | 2 | 3
  >IS 5 | 1 | 5
  >IS 6 | 3 | 3
  >IS 7 | 1 | 9
  >IS+5ASA 1 | 8 | 8
  >IS+5ASA 2 | 15 | 9
  >IS+5ASA 3 | 22 | 10
  >IS+5ASA 4 | 6 | 7
  >IS+5ASA 5 | 3 | 3
  >IS+5ASA 6 | 8 | 5
  >IS+5ASA 7 | 22 | 9
  >No IBD Therapy (NO TR) 1 | 69 | 54
  >NO TR 2 | 217 | 76
  >NO TR 3 | 8 | 0
  >Steroids (STER) 1 | 45 | 35
  >STER 2 | 95 | 28
  >STER 3 | 13 | 14
  >STER 4 | 14 | 6
  >STER 5 | 8 | 2
  Pattern with combination of biologics (BIO COMB) | 35 | 44
  Vedolizumab | 58 | 57
  Other | 22 | 19

2. Secondary Outcome: Number of Participants Stratified by Location of Disease
Time Frame: Within 1 year prior to Baseline (Visit 1)
Population: FAS included those participants who signed the informed consent form and were analyzed in the study. Here, overall number of participants analyzed signified participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1214 | 664
Participants
  Lining of the Rectum | 107 | 0
  Left Side of Colon | 623 | 0
  Ileum | 0 | 146
  Colon | 750 | 183
  Ileum and Colon | 0 | 331
  Upper Gastrointestinal Tract | 0 | 4

3. Secondary Outcome: Number of Participants Stratified by Disease Severity
Description: Disease Severity was defined using Harvey-Bradshaw Index (HBI) and mayo index. HBI is validated clinical index for evaluation of CD disease severity, including the 5 categories: general well-being, abdominal pain, number of liquid stools, abdominal mass and complications. The score ranges from 0 to 25, where score less than (<) 5 was remission, score 5-7 was mild activity, score 8-16 was moderate, and score >16 was severe. Mayo index was used for evaluation of UC disease severity. Mayo index is an instrument consisting of 4 categories of: stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment, each sub score graded from 0 to 3. The score ranges from 0 to 12, where score <2 was remission, score 3-5 was mild, score 6-10 was moderate, and score >10 was severe.
Time Frame: At Visit 1 (Baseline), Visit 2 (6 months), Visit 3 (12 months) of prospective period
Population: FAS included those participants who signed the informed consent form and were analyzed in the study. Here, overall number of participants analyzed signified participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable at specified visits.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1153 | 640
Participants
  Visit 1: Remission | 211 | 322
  Visit 1: Mild | 406 | 166
  Visit 1: Moderate | 522 | 144
  Visit 1: Severe | 14 | 8
  Visit 2: Remission: number analyzed (Participants) | 984 | 502
  Visit 2: Remission | 576 | 339
  Visit 2: Mild: number analyzed (Participants) | 984 | 502
  Visit 2: Mild | 300 | 119
  Visit 2: Moderate: number analyzed (Participants) | 984 | 502
  Visit 2: Moderate | 105 | 43
  Visit 2: Severe: number analyzed (Participants) | 984 | 502
  Visit 2: Severe | 3 | 1
  Visit 3: Remission: number analyzed (Participants) | 945 | 500
  Visit 3: Remission | 614 | 361
  Visit 3: Mild: number analyzed (Participants) | 945 | 500
  Visit 3: Mild | 250 | 103
  Visit 3: Moderate: number analyzed (Participants) | 945 | 500
  Visit 3: Moderate | 81 | 34
  Visit 3: Severe: number analyzed (Participants) | 945 | 500
  Visit 3: Severe | 0 | 2

4. Secondary Outcome: Number of Participants Based on Usage of Methods for Documentation of Disease Activity in Routine Practice
Description: Disease activity assessment was performed using following methods- biomarkers, endoscopy, biopsy, X-ray, magnetic resonance imaging (MRI) and ultrasound examination. Number of participants whose disease activity was evaluated using the respective methods were reported.
Time Frame: From Baseline Visit (Day 1) up to 12 months
Population: FAS included those participants who signed the informed consent form and were analyzed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1214 | 687
Participants
  Biomarkers | 1151 | 662
  Endoscopy | 1188 | 656
  Biopsy | 901 | 453
  X-ray Examination | 206 | 239
  MRI Examination | 138 | 369
  Ultrasound Examination | 283 | 254

5. Secondary Outcome: Number of Assessments Using Different Methods in Participants With UC and CD Disease Activity
Description: Disease activity assessment was performed using following methods- biomarkers, endoscopy, biopsy, X-ray, MRI and ultrasound examination. Biomarkers was based on evaluation of C-reactive protein (CRP) and/or fecal calprotectin levels. Endoscopy included colonoscopy/rectoromanoscopy/sigmoidoscopy and/or video capsule endoscopy and/or esophagogastroduodenoscopy (in the presence or suspicion of the presence of lesions of the upper gastrointestinal tract in Crohn's disease), X-ray was used for examination of the intestine to exclude stricturing and other lesions, MRI was used for examination of the intestine to exclude stricturing and other lesions using MRI and ultrasound for examination of the intestine to exclude stricturing and other lesions. Number of assessments using different methods in participants with UC and CD disease activity was summarized for specified methods and reported in terms of mean and standard deviation.
Time Frame: From Baseline Visit (Day 1) up to 12 months
Population: FAS included those participants who signed the informed consent form and were analyzed in the study.
Measure: Mean (Standard Deviation); unit: assessments
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1214 | 687
assessments
  Biomarkers | 4.52 (4.88) | 6.74 (7.11)
  Endoscopy | 2.60 (1.57) | 2.31 (1.39)
  Biopsy | 1.38 (1.24) | 1.11 (1.16)
  X-ray Examination | 0.23 (0.59) | 0.62 (1.13)
  MRI Examination | 0.15 (0.46) | 1.10 (1.44)
  Ultrasound Examination | 0.53 (1.32) | 1.10 (1.95)

6. Secondary Outcome: UC Participants: Percentage of Participants Who Achieved Combined Clinical and Endoscopic Remission Based on Mayo Index
Description: The full Mayo index is an instrument to measure disease activity of UC. It consists of 4 parameters: stool frequency, rectal bleeding, endoscopic evaluation, and Physician's global assessment. Each parameter of the score ranged from 0 (normal or inactive disease) to 3 (severe activity). The score ranged from 0 to 12, where score <2 was remission, score 3-5 was mild activity, score 6-10 was moderate activity, and score >10 was severe activity. Higher scores indicating higher disease activity.
Time Frame: At Visit 1 (Baseline), Visit 2 (6 months), Visit 3 (12 months) of prospective period
Population: FAS included those participants who signed the informed consent form and were analyzed in the study.
Measure: Number; unit: percentage of participants
Arm/Group | UC Participants
Number analyzed (Participants) | 1214
percentage of participants
  Visit 1: Remission | 18.30
  Visit 1: Mild Activity | 35.21
  Visit 1: Moderate Activity | 45.27
  Visit 1: Severe Activity | 1.21
  Visit 2: Remission | 58.54
  Visit 2: Mild Activity | 30.49
  Visit 2: Moderate Activity | 10.67
  Visit 2: Severe Activity | 0.30
  Visit 3: Remission | 64.97
  Visit 3: Mild Activity | 26.46
  Visit 3: Moderate Activity | 8.57
  Visit 3: Severe Activity | 0.00

7. Secondary Outcome: CD Participants: Percentage of Participants Who Achieved Clinical Remission Based on HBI
Description: HBI was used for evaluation of CD remission. It is a validated clinical index for CD, including the 5 categories of: general well-being, abdominal pain, number of liquid stools, abdominal mass and complications. The score ranges from 0 to 25, where score <5 was remission, score 5-7 was mild activity, score 8-16 was moderate activity, and score >16 was severe activity. Higher scores indicating higher disease activity.
Time Frame: At Visit 1 (Baseline), Visit 2 (6 months), Visit 3 (12 months) of prospective period
Population: FAS included those participants who signed the informed consent form and were analyzed in the study.
Measure: Number; unit: percentage of participants
Arm/Group | CD Participants
Number analyzed (Participants) | 687
percentage of participants
  Visit 1: Remission | 50.31
  Visit 1: Mild Activity | 25.94
  Visit 1: Moderate Activity | 22.50
  Visit 1: Severe Activity | 1.25
  Visit 2: Remission | 67.53
  Visit 2: Mild Activity | 23.71
  Visit 2: Moderate Activity | 8.57
  Visit 2: Severe Activity | 0.20
  Visit 3: Remission | 72.20
  Visit 3: Mild Activity | 20.60
  Visit 3: Moderate Activity | 6.80
  Visit 3: Severe Activity | 0.40

8. Secondary Outcome: Number of Participants With at Least One Episode of Failure of Biological or Non-biological Therapy
Time Frame: From 2 years before enrollment up to Month 12 after enrollment (up to 3 years)
Population: FAS included those participants who signed the informed consent form and were analyzed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1214 | 687
Participants | 1203 | 670

9. Secondary Outcome: Number of Participants Who Needed Treatment Adjustments Based on Disease Activity Assessment
Time Frame: From 2 years before enrollment up to Month 12 after enrollment (up to 3 years)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 35 | 35
Participants
  If an Exacerbation or Deterioration Developed | 0 [lower limit 15.0] | 1 [lower limit 21.0]
  Every 3 months, as well as in the Development of Exacerbation or Deterioration | 14 [lower limit 19.2] | 10 [lower limit 22.0]
  Every six months, as well as When the Exacerbation or Deterioration | 11 [lower limit 21.4] | 15 [lower limit 22.4]
  Once a year, as well as in the Case of the Development of Exacerbation or Deteriorations | 9 [lower limit 23.7] | 8 [lower limit 24.4]

10. Secondary Outcome: Percentage of Participants Stratified by Achieving the Treatment Goals
Description: Treat to target (T2T) approach was used for assessment of treatment goals. A "Treat to target" approach for UC included clinical remission (defined as resolution of rectal bleeding and diarrhea/altered bowel habit) and endoscopic remission (defined as Mayo endoscopic subscore of 0-1). Biomarker remission (normal C-reactive protein [CRP] and calprotectin) was considered as an adjunctive target. Histological remission was considered as an adjunctive goal. Clinical remission for CD was defined as resolution of abdominal pain and diarrhea/altered bowel habit. Endoscopic remission for CD was defined as resolution of ulceration at ileocolonoscopy or resolution of findings of inflammation on cross-sectional imaging in participants who cannot be adequately assessed with ileocolonoscopy. Biomarker remission (normal CRP and faecal calprotectin) was considered as an adjunctive target.
Time Frame: From 2 years before enrollment up to Month 12 after enrollment (up to 3 years)
Population: FAS included those participants who signed the informed consent form and were analyzed in the study. Here, overall number of participants analyzed signified participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for given categories.
Measure: Number; unit: percentage of participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 35 | 35
percentage of participants
  Clinical Remission: number analyzed (Participants) | 34 | 34
  Clinical Remission | 81.3 | 70.3
  Endoscopic Remission: number analyzed (Participants) | 34 | 34
  Endoscopic Remission | 61.2 | 50.6
  Histological Remission: number analyzed (Participants) | 30 | 28
  Histological Remission | 29.8 | 27.4
  Biomarker Remission: number analyzed (Participants) | 31 | 32
  Biomarker Remission | 75.9 | 68.1

11. Secondary Outcome: Percentage of Participants Based on Challenges of Implementing a T2T Strategy in UC and CD Participants in Real Clinical Practice
Description: "Other" challenges included absence or inaccessibility of MRI (technical problems), participants financial difficulties, disability and bureaucratic problems, unavailability of biotherapy, limited quotas, referral of participants to other centers, absence of biotherapy treatment quotas, difficulty in performing computed tomography (CT).
Time Frame: From 2 years before enrollment up to Month 12 after enrollment (up to 3 years)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 35 | 35
percentage of participants
  Difficulties or Inaccessibility of Colonoscopy | 28.6 | 28.6
  Unwillingness to Undergo Colonoscopy | 40.0 | 45.7
  Participant's Failure to Follow Visit Scheduled With Physician | 40.0 | 40.0
  Participant's Non-compliance With Drug Therapy | 45.7 | 51.4
  Resistant Course of Disease | 71.4 | 71.4
  Difficulties or Unavailability of Certain Drugs | 65.7 | 57.1
  Workload of Doctor | 28.6 | 22.9
  Lack of Participants Record System and Monitoring | 25.7 | 22.9
  Other | 14.3 | 20.0

12. Secondary Outcome: Percentage of Participants Based on Hospitalizations Due to Complications, IBD Related Surgeries, and Disability Determination in Participants With Moderate to Severe UC and CD
Time Frame: From 2 years before enrollment up to Month 12 after enrollment (up to 3 years)
Population: FAS included those participants who signed the informed consent form and were analyzed in the study.
Measure: Number; unit: percentage of participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1214 | 687
percentage of participants
  Hospitalizations due to Complications | 2.14 | 3.06
  IBD Related Surgeries | 0.33 | 0.73
  IBD Related Disability | 29.57 | 47.74

13. Secondary Outcome: Percentage of Participants Based on Surgical Treatment by Indications and Type of Surgeries
Description: Indications for surgical treatment included aggravation, intestinal bleeding, colon perforation, internal fistulas, abdominal cavity infiltrate, Interintestinal or Intraabdominal abscess, strictures in the gastrointestinal tract, anal fissures, and other. Types of surgeries includes both emergency and planned.
Time Frame: From 2 years before enrollment up to Month 12 after enrollment (up to 3 years)
Population: FAS included those participants who signed the informed consent form and were analyzed in the study. Here, number analyzed signifies participants who were evaluable for given categories.
Measure: Number; unit: percentage of participants
Arm/Group | UC Participants | CD Participants
Number analyzed (Participants) | 1214 | 687
percentage of participants
  Surgical Treatment by Indication: Aggravation | 0.58 | 0.58
  Surgical Treatment by Indication: Intestinal Bleeding: number analyzed (Participants) | 1214 | 0
  Surgical Treatment by Indication: Intestinal Bleeding | 0.49 |
  Surgical Treatment by Indication: Colon Perforation | 0.08 | 0.15
  Surgical Treatment by Indication: Other | 0.99 | 1.16
  Surgical Treatment by Indication: Internal Fistulas: number analyzed (Participants) | 0 | 687
  Surgical Treatment by Indication: Internal Fistulas |  | 0.15
  Surgical Treatment by Indication: Abdominal Cavity Infiltrate: number analyzed (Participants) | 0 | 687
  Surgical Treatment by Indication: Abdominal Cavity Infiltrate |  | 0.15
  Surgical Treatment by Indication: Interintestinal or Intraabdominal Abscess: number analyzed (Participants) | 0 | 687
  Surgical Treatment by Indication: Interintestinal or Intraabdominal Abscess |  | 0.29
  Surgical Treatment by Indication: Strictures in the gastrointestinal tract: number analyzed (Participants) | 0 | 687
  Surgical Treatment by Indication: Strictures in the gastrointestinal tract |  | 1.16
  Surgical Treatment by Indication: Anal Fissures: number analyzed (Participants) | 0 | 687
  Surgical Treatment by Indication: Anal Fissures |  | 0.15
  Type of Surgeries: Emergency | 0.16 | 0.29
  Type of Surgeries: Planned | 0.25 | 0.58

ADVERSE EVENTS:
Time Frame: Up to 12 months after enrollment into the study
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety data was not planned to be collected for this observational retrospective part of the study, however it was collected and assessed for the prospective part of the study.
Arm/Group | UC Participants | CD Participants
All-Cause Mortality (participants affected / at risk) | 3/1214 | 5/687
Serious Adverse Events (participants affected / at risk) | 146/1214 | 84/687
Other Adverse Events (participants affected / at risk) | 48/1214 | 31/687
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UC Participants (N=1214) | CD Participants (N=687)
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 124 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 1 | 0
Acute hepatitis C (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Cervical leukoplakia (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colitis ulcerative (Surgical and medical procedures) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 56
Ileal stenosis (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Intestinal stenosis (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Enterocolonic fistula (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Small intestinal resection (Surgical and medical procedures) | 0 | 1
Ileectomy (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Takayasu's arteritis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UC Participants (N=1214) | CD Participants (N=687)
Leukopenia (Blood and lymphatic system disorders) | 7 | 5
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 4 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Drug resistance (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Loss of therapeutic response (General disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 2
Bartholin's abscess (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0
Transaminases increased (Investigations) | 3 | 2
Cell death (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Cervical leukoplakia (Reproductive system and breast disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Abscess drainage (Surgical and medical procedures) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Drug ineffective (General disorders) | 0 | 1
Loss of therapeutic response (General disorders) | 0 | 1
Drug induced liver injury (Hepatobiliary disorders) | 1 | 3
Drug hypersensitivity (Immune system disorders) | 2 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia totalis (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT03532932/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT03532932/SAP_001.pdf